CLINICAL TRIAL: NCT06124729
Title: Evaluation of the Efficacy and Safety of Bevacizumab Combined With PD-1 Monoclonal Antibody in Preoperative Neoadjuvant Therapy for MSS Colorectal Cancer With Liver Metastases - a Single-center, Single-arm, Open-label Clinical Trail
Brief Title: Evaluation of the Efficacy and Safety of Bevacizumab Combined With PD-1 Monoclonal Antibody in Preoperative Neoadjuvant Therapy for MSS Colorectal Cancer With Liver Metastases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: CRSYM202311
Record Dates: First submitted 2023-11-05; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Bevacizumab Combined With PD-1 Monoclonal Antibody in Preoperative Neoadjuvant Therapy
  Interventions: Drug: Bevacizumab Combined With PD-1 Monoclonal Antibody

INTERVENTIONS:
Drug: Bevacizumab Combined With PD-1 Monoclonal Antibody — Bevacizumab Combined With PD-1 Monoclonal Antibody in Preoperative Neoadjuvant Therapy for MSS colorectal cancer with liver metastases

SUMMARY:
Evaluation of the Efficacy and Safety of Bevacizumab Combined With PD-1 Monoclonal Antibody in Preoperative Neoadjuvant Therapy for MSS Colorectal Cancer With Liver Metastases - a Single-center, Single-arm, Open-label Clinical Trail.

DETAILED DESCRIPTION:
In the 2023 Global Cancer Statistics, colorectal cancer remains the third leading cause of cancer-related death in the world. According to the latest China Cancer report, colorectal cancer is the fourth leading cause of cancer-related death in China. More specifically, the incidence and the mortality of colorectal cancer have been increasing year over year. Among newly diagnosed colorectal cancer patients, 20% have distant metastases. The 5-year survival rate for metastatic colorectal cancer (mCRC) is less than 20%. In the latest updated 2023 National Cancer Comprehensive Network (NCCN) Colon Cancer Guidelines, mismatch repair genes/micro satellite state officially became a global classification standard. Patients diagnosed with colorectal cancer must be classified into MSS or MSI-H before treatment, that is, patients are divided into pMMR/MSS and dMMR/MSI-H subtypes after initial examination or clinical management, and then the treatment plan is determined. MSI-H accounts for 15% of all colorectal cancers and is mostly present in patients with early stage tumors. For patients with metastatic colorectal cancer, MSI-H colorectal cancer accounts for only 5% of all patients. Among them, the treatment of immune checkpoint inhibitors in MSI-H patients has become a first-line and neoadjuvant metastatic disease treatment recommendation.

Although clinical trials on the combination of targeted therapy and immunotherapy are increasing, clinical researches and clinical trials of targeted therapy combined immunotherapy, such as bevacizumab combined with PD-1, have not received enough attention and recognition. Currently reports believed that anti-programmed death-1 (PD-1) antibodies have been shown to produce significantly longer progression-free survival with fewer adverse events compared to chemotherapy as a first-line treatment for dMMR metastatic CRC (mCRC). In the simultaneous CRT sequential PD-1 (long range) and TNT simultaneous combined PD-1 (long range) clinical trials, CRT combined with PD-1/PD-L1 showed better near-term efficacy gains (pCR) in patients with locally staged pMMR. Although current researches on neoadjuvant therapy for MSS type bowel cancer is increasingly abundant, especially PD-1 is becoming more and more popular in the treatment of MSS type bowel cancer, the research in the field of neoadjuvant therapy for MSS metastatic colorectal cancer is still not explored. Therefore, our PD-1 combined with bevacizumab in the treatment of MSS type metastatic bowel cancer has greatly research value.

Based on the above reasons, we designed this study to observe the efficacy and safety of the target-free combination therapy regimen of PD-1 combined with bevacizumab for patients with MSS metastatic colorectal cancer, and strive to provide a high-level evidence-based basis for neoadjuvant therapy regimen for patients with MSS metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-75 years old;
2. Histologically or radiographically proven colon or rectal adenocarcinoma with liver metastases；
3. ECOG performance status score of 0 to 2；
4. Clinical staged any T with liver metastases (M+);
5. MSS status;
6. Adequate haematological, hepatic, and renal function: neutrophil count ≥1.5×109 /L; platelet count ≥75×109 /L; serum total bilirubin ≤1.5×upper normal limits (UNL); aspartate aminotransferase ≤2.5×UNL; alanine aminotransferase ≤2.5×UNL; serum creatinine ≤1.5 x UNL.

Exclusion Criteria:

1. MSI status;
2. Colorectal cancer without liver metastases;
3. Relapsed colorectal cancer;
4. Complicated with active bleeding, perforation, or requiring emergency surgery;
5. Previous systemic anticancer therapy for colorectal cancer disease;
6. Any active or history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications;
7. Patients with other active concurrent non-colorectal cancer;
8. Patients with interstitial lung disease, non-infectious pneumonia or uncontrollable systemic diseases (such as: diabetes, hypertension, pulmonary fibrosis and acute pneumonia);
9. Patients with any Grade 2 or above toxicity as classified by the common terminology criteria for adverse events (CTCAE) (version 5.0) (except for anemia, alopecia and skin pigmentation) which is induced by previous treatment and has not subside;
10. Previously received anti-programmed death-1 (PD-1) or its ligand (PD-L1) antibody, anti- cytotoxic T lymphocyte-associated antigen 4 (cytotoxic T-lymphocyte-associated Protein 4, CTLA-4) antibody Women in pregnancy or lactation;
11. Known positive history or positive test for Human Immunodeficiency Virus or Acquired Immunodeficiency Syndrome (AIDS);
12. History of known or suspected allergies to any related drugs used in the trial; Women who are pregnant or nursing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MSS colorectal cancer who have been diagnosed with liver metastases and are physically able to tolerate neoadjuvant chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
cCR | 20 weeks
  To evaluate whether neoadjuvant Bevacizumab Combined With PD-1 Monoclonal Antibody would significantly improve the Clinical complete response (cCR) proportion in MSS Colorectal Cancer With Liver Metastases

SECONDARY OUTCOMES:
R0 resection rate | 1 day
  To evaluate whether neoadjuvant Bevacizumab Combined With PD-1 Monoclonal Antibody would significantly improve the R0 resection rate in MSS Colorectal Cancer With Liver Metastases
pCR proportion | 20 weeks
  To evaluate whether neoadjuvant Bevacizumab Combined With PD-1 Monoclonal Antibody would significantly improve the pCR proportion in MSS Colorectal Cancer With Liver Metastases
Major pathological response (MPR) | 20 weeks
  To evaluate whether neoadjuvant Bevacizumab Combined With PD-1 Monoclonal Antibody would significantly improve the Major pathological response proportion in MSS Colorectal Cancer With Liver Metastases
Disease-free survival (DFS) and overall survival (OS) | 5 years
  To evaluate whether neoadjuvant Bevacizumab Combined With PD-1 Monoclonal Antibody would significantly improve the RFS and OS rate in MSS Colorectal Cancer With Liver Metastases

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diaz LA Jr, Shiu KK, Kim TW, Jensen BV, Jensen LH, Punt C, Smith D, Garcia-Carbonero R, Benavides M, Gibbs P, de la Fourchardiere C, Rivera F, Elez E, Le DT, Yoshino T, Zhong WY, Fogelman D, Marinello P, Andre T; KEYNOTE-177 Investigators. Pembrolizumab versus chemotherapy for microsatellite instability-high or mismatch repair-deficient metastatic colorectal cancer (KEYNOTE-177): final analysis of a randomised, open-label, phase 3 study. Lancet Oncol. 2022 May;23(5):659-670. doi: 10.1016/S1470-2045(22)00197-8. Epub 2022 Apr 12. PMID 35427471